CLINICAL TRIAL: NCT01395849
Title: Drug Use Investigation for ADOAIR (Fluticasone/Salmeterol)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112277
Record Dates: First submitted 2011-07-14; First posted 2011-07-18 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Respiratory Disorders
MeSH Terms: conditions — Respiration Disorders | interventions — Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients prescribed fluticasone and salmeterol: Patients with asthma prescribed fluticasone and salmeterol during study period
  Interventions: Drug: Salmeterol and Fluticasone

INTERVENTIONS:
Drug: Salmeterol and Fluticasone

SUMMARY:
The purpose of this post-marketing surveillance is to detect adverse drug reactions (particularly clinically significant adverse drug reactions) occurring in clinical settings, to examine factors likely to affect the safety and efficacy in the Japanese asthma patients treated with fluticasone propionate and salmeterol xinafoate.

ELIGIBILITY:
Inclusion Criteria:

* Must use fluticasone and salmeterol for the first time

Exclusion Criteria:

* Patients with hypersensitivity to salmeterol and fluticasone
* Patients with infection which salmeterol and fluticasone is not effective
* Patients with deep mycosis

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Japanese patients with asthma
Sampling Method: Probability Sample
Enrollment: 2116 (Actual)
Dates: Start 2007-10; Primary Completion 2009-09 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The number of incidence of adverse events in Japanese asthma patients treated with fluticasone propionate and salmeterol xinafoate | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline